CLINICAL TRIAL: NCT05051241
Title: A Phase I Study With Single/Multiple Dose Administered to Explore the Safety/Tolerability and Pharmacokinetics of GFH018 in the Treatment of Patients With Advanced Solid Tumors
Brief Title: A Study of GFH018 in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zhejiang Genfleet Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Genfleet Therapeutics (Shanghai) Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GFH018X1101
Record Dates: First submitted 2021-09-02; First posted 2021-09-21 (Actual); Results first posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2023-07

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Dose escalation Cohort 1 (Experimental): 5 mg BID, 14d-on/14d-off
  Interventions: Drug: GFH018
- Dose escalation Cohort 2 (Experimental): 10 mg BID, 14d-on/14d-off
  Interventions: Drug: GFH018
- Dose escalation Cohort 3 (Experimental): 20 mg BID, 14d-on/14d-off
  Interventions: Drug: GFH018
- Dose escalation Cohort 4 (Experimental): 30 mg BID, 14d-on/14d-off
  Interventions: Drug: GFH018
- Dose escalation Cohort 5 (Experimental): 40 mg BID, 14d-on/14d-off
  Interventions: Drug: GFH018
- Dose escalation Cohort 6 (Experimental): 50 mg BID, 14d-on/14d-off
  Interventions: Drug: GFH018
- Dose escalation Cohort 7 (Experimental): 65 mg BID, 14d-on/14d-off
  Interventions: Drug: GFH018
- Dose escalation Cohort 8 (Experimental): 85 mg BID, 14d-on/14d-off
  Interventions: Drug: GFH018
- Dose escalation Cohort 9 (Experimental): 85 mg BID, 7d-on/7d-off
  Interventions: Drug: GFH018
- Dose expansion Cohort 10 (Experimental): 85 mg BID, 14d-on/14d-off
  Interventions: Drug: GFH018

INTERVENTIONS:
Drug: GFH018 — Subjects will receive GFH018 orally at different dose levels following twice daily, 14-day on/14-day off regimen. Other dose regimens, eg 7d-on/7d-off will also be considered to be explored when the safety/tolerability is confirmed.

SUMMARY:
This is the first- in human study of GFH018 comprised of a dose escalation part and a dose expansion part in subjects with advanced solid tumors after single/multiple administration. The study is designed to explore the safety/tolerability, pharmacokinetics, and MTD of GFH018 and to define a RP2D of GFH018.

ELIGIBILITY:
Inclusion Criteria:

* Eligible subjects must meet all the inclusion criteria listed below:

  1. Voluntarily participate in this clinical trial and are willing to sign informed consent forms.
  2. Male or female aged from 18-75 years old (inclusive).
  3. Diagnosed with histologically or cytologically confirmed advanced solid tumors.
  4. Evaluable lesions defined by RECIST v1.1.
  5. Eastern Cooperative Oncology Group performance status of 0 to 1.
  6. Subjects or their legal representatives are able to communicate well with Investigators and are willing to comply with the protocol and complete the study.

Exclusion Criteria:

* Eligible subjects should not meet any of the exclusion criteria listed below:

  1. With clinically significant cardiac diseases.
  2. With clinically significant digestive disorders.
  3. Other severe disease.
  4. Pregnant or lactating women.
  5. Other unfavorable situations for subjects to participate in the study judged by Investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-08-30 (Actual); Primary Completion 2022-08-11 (Actual); Study Completion 2022-08-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, MD, Principal Investigator — Leading site
Locations (1):
- Shanghai East hospital, Shanghai, China

REFERENCES:
- [Derived] Guo Y, Wang Z, Zhou H, Pan H, Han W, Deng Y, Li Q, Xue J, Ge X, Wang S, Wang J, Zhang Y, Zhao C, Zhu H, Wang Y, Shen H, Liu D, Li J. First-in-human study of GFH018, a small molecule inhibitor of transforming growth factor-beta receptor I inhibitor, in patients with advanced solid tumors. BMC Cancer. 2024 Apr 10;24(1):444. doi: 10.1186/s12885-024-12216-7. PMID 38600507

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 50 participants who met all inclusion and no exclusion criteria were enrolled at 5 centers in China. A total of 47 participants started the Dose Escalation phase and three participants in the Dose Expansion phase.
Pre-assignment Details: The Dose Escalation was intended to identify the maximum tolerated dose (MTD) or recommended phase 2 dose (RP2D) of GFH018 with at least 3 participants evaluable for assessment of dose-limiting toxicity per dose level. Since the MTD was not reached, 85 mg BID, 14d-on/14d-off was chosen for evaluation in the Dose Expansion phase.
Groups:
- Dose Escalation: Cohort 1 5 mg BID, 14d-on/14d-off: Participants in Cohort 1 received GFH018 5 mg BID, 14d-on/14d-off orally
- Dose Escalation: Cohort 2 10 mg BID, 14d-on/14d-off: Participants in Cohort 2 received GFH018 10 mg BID, 14d-on/14d-off
- Dose Escalation: Cohort 3 20 mg BID, 14d-on/14d-off: Participants in Cohort 3 received GFH018 20 mg BID, 14d-on/14d-off
- Dose Escalation: Cohort 4 30 mg BID, 14d-on/14d-off: Participants in Cohort 4 received GFH018 30 mg BID, 14d-on/14d-off orally
- Dose Escalation: Cohort 5 40 mg BID, 14d-on/14d-off: Participants in Cohort 5 received GFH018 40 mg BID, 14d-on/14d-off orally
- Dose Escalation: Cohort 6 50 mg BID, 14d-on/14d-off: Participants in Cohort 6 received GFH018 50 mg BID, 14d-on/14d-off orally
- Dose Escalation: Cohort 7 65 mg BID, 14d-on/14d-off: Participants in Cohort 7 received GFH018 65 mg BID, 14d-on/14d-off orally
- Dose Escalation: Cohort 8 85 mg BID, 14d-on/14d-off: Participants in Cohort 8 received GFH018 85 mg BID, 14d-on/14d-off orally
- Dose Escalation: Cohort 9 85 mg BID, 7d-on/7d-off: Participants in Cohort 9 received GFH018 85 mg BID, 7d-on/7d-off orally
- Dose Expansion: Cohort 10 85 mg BID, 14d-on/14d-off: Participants in Cohort 10 received GFH018 85 mg BID, 14d-on/14d-off orally
Period: Dose Escalation
Arm/Group | Dose Escalation: Cohort 1 5 mg BID, 14d-on/14d-off | Dose Escalation: Cohort 2 10 mg BID, 14d-on/14d-off | Dose Escalation: Cohort 3 20 mg BID, 14d-on/14d-off | Dose Escalation: Cohort 4 30 mg BID, 14d-on/14d-off | Dose Escalation: Cohort 5 40 mg BID, 14d-on/14d-off | Dose Escalation: Cohort 6 50 mg BID, 14d-on/14d-off | Dose Escalation: Cohort 7 65 mg BID, 14d-on/14d-off | Dose Escalation: Cohort 8 85 mg BID, 14d-on/14d-off | Dose Escalation: Cohort 9 85 mg BID, 7d-on/7d-off | Dose Expansion: Cohort 10 85 mg BID, 14d-on/14d-off
Started | 4 | 3 | 4 | 7 | 4 | 4 | 6 | 9 | 6 | 0
Completed | 4 | 3 | 4 | 7 | 4 | 4 | 6 | 9 | 6 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Dose Expansion
Arm/Group | Dose Escalation: Cohort 1 5 mg BID, 14d-on/14d-off | Dose Escalation: Cohort 2 10 mg BID, 14d-on/14d-off | Dose Escalation: Cohort 3 20 mg BID, 14d-on/14d-off | Dose Escalation: Cohort 4 30 mg BID, 14d-on/14d-off | Dose Escalation: Cohort 5 40 mg BID, 14d-on/14d-off | Dose Escalation: Cohort 6 50 mg BID, 14d-on/14d-off | Dose Escalation: Cohort 7 65 mg BID, 14d-on/14d-off | Dose Escalation: Cohort 8 85 mg BID, 14d-on/14d-off | Dose Escalation: Cohort 9 85 mg BID, 7d-on/7d-off | Dose Expansion: Cohort 10 85 mg BID, 14d-on/14d-off
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dose Escalation Cohort 1 5 mg BID, 14d-on/14d-off: Participants in Cohort 1 received GFH018 5 mg BID, 14d-on/14d-off orally
- Dose Escalation: Cohort 4 30 mg BID, 14d-on/14d-off: Participants in Cohort 4 received GFH018 30 mg BID, 14d-on/14d-off
- Dose Escalation: Cohort 5 40 mg BID, 14d-on/14d-off: Participants in Cohort 5 received GFH018 40 mg BID, 14d-on/14d-off
- Dose Escalation: Cohort 6 50 mg BID, 14d-on/14d-off: Participants in Cohort 6 received GFH018 50 mg BID, 14d-on/14d-off
- Dose Escalation: Cohort 7 65 mg BID, 14d-on/14d-off: Participants in Cohort 7 received GFH018 65 mg BID, 14d-on/14d-off
- Dose Escalation: Cohort 8 85 mg BID, 14d-on/14d-off: Participants in Cohort 8 received GFH018 85 mg BID, 14d-on/14d-off
- Dose Escalation: Cohort 9 85 mg BID, 7d-on/7d-off: Participants in Cohort 9 received GFH018 85 mg BID, 7d-on/7d-off
- Dose Expansion: Cohort 10 85 mg BID, 14d-on/14d-off: Participants in Cohort 10 received GFH018 85 mg BID, 14d-on/14d-off
- Total: Total of all reporting groups
Arm/Group | Dose Escalation Cohort 1 5 mg BID, 14d-on/14d-off | Dose Escalation: Cohort 2 10 mg BID, 14d-on/14d-off | Dose Escalation: Cohort 3 20 mg BID, 14d-on/14d-off | Dose Escalation: Cohort 4 30 mg BID, 14d-on/14d-off | Dose Escalation: Cohort 5 40 mg BID, 14d-on/14d-off | Dose Escalation: Cohort 6 50 mg BID, 14d-on/14d-off | Dose Escalation: Cohort 7 65 mg BID, 14d-on/14d-off | Dose Escalation: Cohort 8 85 mg BID, 14d-on/14d-off | Dose Escalation: Cohort 9 85 mg BID, 7d-on/7d-off | Dose Expansion: Cohort 10 85 mg BID, 14d-on/14d-off | Total
Number analyzed (Participants) | 4 | 3 | 4 | 7 | 4 | 4 | 6 | 9 | 6 | 3 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 3 | 6 | 4 | 4 | 6 | 8 | 5 | 3 | 44
  >=65 years | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 6
Age, Continuous [Median (Full Range); unit: years] | 53.5 [40 to 67] | 39 [27 to 68] | 50.5 [39 to 67] | 51 [40 to 66] | 51.5 [44 to 60] | 55 [36 to 61] | 56.5 [34 to 63] | 52 [39 to 67] | 52.5 [47 to 66] | 49 [47 to 55] | 52.5 [27 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3 | 3 | 3 | 1 | 5 | 5 | 2 | 2 | 27
  Male | 3 | 1 | 1 | 4 | 1 | 3 | 1 | 4 | 4 | 1 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 4 | 3 | 4 | 7 | 4 | 4 | 6 | 9 | 6 | 3 | 50
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 4 | 3 | 4 | 7 | 4 | 4 | 6 | 9 | 6 | 3 | 50

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Dose-limiting Toxicity (DLT) Events
Time Frame: 31 days after the first dose
Population: Participants enrolled in the expansion part were NOT included in analyzing the incidence of DLT. So the analyzed number of cohort 10 was 0.
Measure: Count of Participants; unit: Participants
Groups:
- Dose Escalation: Cohort 2 10 mg BID, 14d-on/14d-off: Participants in Cohort 2 received GFH018 10 mg BID, 14d-on/14d-off orally
- Dose Escalation: Cohort 3 20 mg BID, 14d-on/14d-off: Participants in Cohort 3 received GFH018 20 mg BID, 14d-on/14d-off orally
Arm/Group | Dose Escalation: Cohort 1 5 mg BID, 14d-on/14d-off | Dose Escalation: Cohort 2 10 mg BID, 14d-on/14d-off | Dose Escalation: Cohort 3 20 mg BID, 14d-on/14d-off | Dose Escalation: Cohort 4 30 mg BID, 14d-on/14d-off | Dose Escalation: Cohort 5 40 mg BID, 14d-on/14d-off | Dose Escalation: Cohort 6 50 mg BID, 14d-on/14d-off | Dose Escalation: Cohort 7 65 mg BID, 14d-on/14d-off | Dose Escalation: Cohort 8 85 mg BID, 14d-on/14d-off | Dose Escalation: Cohort 9 85 mg BID, 7d-on/7d-off | Dose Expansion: Cohort 10 85 mg BID, 14d-on/14d-off
Number analyzed (Participants) | 4 | 3 | 4 | 7 | 4 | 4 | 6 | 9 | 6 | 0
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse event (TEAE) data were collected from baseline up to 30 days after the last dose of study drug, up to 1 years.
Description: TEAEs were AEs that occur, having been absent before the first dose of study drug, or has worsened in severity or seriousness after the first dose until 30 days after the last dose. Serious adverse events with an onset or worsening ≥30 days after the last dose, if related to the study treatment, are also TEAEs.
Groups:
- Dose Escalation: Cohort 3 20 mg BID, 14d-on/14d-off: Participants in Cohort 3 received GFH018 10 mg BID, 14d-on/14d-off orally
- Dose Escalation: Cohort 7 65 mg BID, 14d-on/14d-off: Participants in Cohort 7 received GFH01865 mg BID, 14d-on/14d-off orally
- Dose Escalation: Cohort 9 85 mg BID, 7d-on/7d-off: Participants in Cohort 9 received GFH018 85 mg BID, 7d-on/17d-off orally
Arm/Group | Dose Escalation: Cohort 1 5 mg BID, 14d-on/14d-off | Dose Escalation: Cohort 2 10 mg BID, 14d-on/14d-off | Dose Escalation: Cohort 3 20 mg BID, 14d-on/14d-off | Dose Escalation: Cohort 4 30 mg BID, 14d-on/14d-off | Dose Escalation: Cohort 5 40 mg BID, 14d-on/14d-off | Dose Escalation: Cohort 6 50 mg BID, 14d-on/14d-off | Dose Escalation: Cohort 7 65 mg BID, 14d-on/14d-off | Dose Escalation: Cohort 8 85 mg BID, 14d-on/14d-off | Dose Escalation: Cohort 9 85 mg BID, 7d-on/7d-off | Dose Expansion: Cohort 10 85 mg BID, 14d-on/14d-off
All-Cause Mortality (participants affected / at risk) | 1/4 | 0/3 | 0/4 | 2/7 | 0/4 | 0/4 | 0/6 | 2/9 | 1/6 | 0/3
Serious Adverse Events (participants affected / at risk) | 1/4 | 0/3 | 0/4 | 5/7 | 0/4 | 0/4 | 0/6 | 2/9 | 1/6 | 1/3
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3 | 4/4 | 7/7 | 4/4 | 2/4 | 5/6 | 8/9 | 3/6 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation: Cohort 1 5 mg BID, 14d-on/14d-off (N=4) | Dose Escalation: Cohort 2 10 mg BID, 14d-on/14d-off (N=3) | Dose Escalation: Cohort 3 20 mg BID, 14d-on/14d-off (N=4) | Dose Escalation: Cohort 4 30 mg BID, 14d-on/14d-off (N=7) | Dose Escalation: Cohort 5 40 mg BID, 14d-on/14d-off (N=4) | Dose Escalation: Cohort 6 50 mg BID, 14d-on/14d-off (N=4) | Dose Escalation: Cohort 7 65 mg BID, 14d-on/14d-off (N=6) | Dose Escalation: Cohort 8 85 mg BID, 14d-on/14d-off (N=9) | Dose Escalation: Cohort 9 85 mg BID, 7d-on/7d-off (N=6) | Dose Expansion: Cohort 10 85 mg BID, 14d-on/14d-off (N=3)
Sudden death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neoplasma progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proteinuira (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation: Cohort 1 5 mg BID, 14d-on/14d-off (N=4) | Dose Escalation: Cohort 2 10 mg BID, 14d-on/14d-off (N=3) | Dose Escalation: Cohort 3 20 mg BID, 14d-on/14d-off (N=4) | Dose Escalation: Cohort 4 30 mg BID, 14d-on/14d-off (N=7) | Dose Escalation: Cohort 5 40 mg BID, 14d-on/14d-off (N=4) | Dose Escalation: Cohort 6 50 mg BID, 14d-on/14d-off (N=4) | Dose Escalation: Cohort 7 65 mg BID, 14d-on/14d-off (N=6) | Dose Escalation: Cohort 8 85 mg BID, 14d-on/14d-off (N=9) | Dose Escalation: Cohort 9 85 mg BID, 7d-on/7d-off (N=6) | Dose Expansion: Cohort 10 85 mg BID, 14d-on/14d-off (N=3)
AST increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 0 (0)
Lymphocyte count decreased (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
ALT increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urine protein present (Investigations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
GGT increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
ALP increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
LDH increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Electrocardiogram T wave abnormal (Investigations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Peripheral edema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After the completion of the research, researchers can collaborate with the sponsoring party for publication. Researchers must commit not to submit any part of the data from this study for publication without prior approval from the sponsoring party.

DOCUMENTS (2):
  • Study Protocol (2021-03-02): https://cdn.clinicaltrials.gov/large-docs/41/NCT05051241/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-31): https://cdn.clinicaltrials.gov/large-docs/41/NCT05051241/SAP_001.pdf